CLINICAL TRIAL: NCT05452356
Title: Testing of Patient Care Sets and Management of Cardiovascular Conditions Using a Virtual Platform
Brief Title: Testing VIRTUES Patient Care Sets in Cardiac Patients (VIRTUES Cardiac Care)
Acronym: VIRTUES-CC
Status: Recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Cardiac Arrhythmia Network of Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 12505
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-03

CONDITIONS: Heart Diseases; Arrhythmias, Cardiac; Atrial Fibrillation; Cardiovascular Diseases; Pathologic Processes
MeSH Terms: conditions — Heart Diseases; Arrhythmias, Cardiac; Atrial Fibrillation; Cardiovascular Diseases; Pathologic Processes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with various cardiac conditions (such as those who experience a heart attack) are increasing in Canada and are in need of appropriate cardiac rehabilitation and care. Many patients do not have access to local in-person cardiac clinics, particularly in rural regions of Canada. A user-friendly digital application with accessible educational resources and recommendations based on the most up to date clinical practice guidelines can help mitigate these issues. VIRTUES is a digital healthcare application that targets 11 modifiable modules as follows:

1. antithrombotic management
2. lipid management
3. rate and rhythm control for atrial fibrillation
4. heart failure care
5. post myocardial infarction care
6. blood sugar management
7. blood pressure management
8. physical activity
9. healthy eating
10. smoking cessation
11. alcohol reduction

Of the 11 total modules, the first 7 listed provide recommendations in VIRTUES. The remaining 4 (physical activity, healthy eating, smoking cessation and alcohol reduction) consist of simple referrals to existing recommendations (i.e., for healthy eating and physical exercise) and referrals to existing local programs (i.e., for smoking cessation and alcohol reduction). Thus, in this cohort study, the investigators will test the primary 7 modules with 200 patients per module for approximately one month each in order to obtain feedback on the usability of each module. The investigators will also conduct virtual focus group discussions to obtain open ended feedback on the application. This study will provide valuable feedback, which will be used to improve and adapt the VIRTUES platform.

DETAILED DESCRIPTION:
Heart conditions are on the rise in Canada, contributing substantially to patient quality of life. For example, over 60,000 Canadians will experience a heart attack per year. Other conditions, such as Atrial Fibrillation (in which the heart beats rapidly and irregularly) are also highly prevalent, with an estimated 250% increase by 2050. Unfortunately, few patients receive appropriate cardiac rehabilitation, and local in-person cardiac clinics are often inaccessible in rural regions. Patients need user-friendly, accessible educational resources based on current clinical practice guidelines. A digital interphase where patients can access their health information easily, and receive accurate medical advice can significantly help them manage their conditions. VIRTUES ("Virtual Integrated Reliable Transformative User Driven E-Health System") is a digital healthcare platform developed in partnership with the Cardiovascular Network of Canada (CANet). VIRTUES is a web application that uses built-in algorithms specific to each patient to make guideline-directed recommendations to patients and their healthcare providers and provide individually tailored educational material. VIRTUES includes the following 11 targeted modules:

1. antithrombotic management
2. lipid management
3. rate and rhythm control for atrial fibrillation
4. heart failure care
5. post myocardial infarction care
6. blood sugar management
7. blood pressure management
8. physical activity
9. healthy eating
10. smoking cessation
11. alcohol reduction

Of the 11 total modules, the first 7 listed provide recommendations to patients in VIRTUES. The remaining 4 (physical activity, healthy eating, smoking cessation and alcohol reduction) consist of simple referrals to existing local programs. The current cohort study tests the feasibility, usability, and patient experience of using VIRTUES in 200 patients across the 7 targeted modules that provide individually tailored recommendations. Each patient will only be exposed to module(s) specific to her/his condition. Testing will take place over the duration of approximately one month per module with approximately 1,400 patients in total (200 patients enrolled in each of the 7 modules). Patients will complete a series of forms assessing their medical history at the beginning of the study and they will be given a survey on their experience using VIRTUES after 6 and 12 months of using it. Patients will also be given an opportunity to volunteer for a virtual focus group discussion with other patients. The goal of this study is to provide insights on how to modify and improve VIRTUES based on patient feedback.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a cardiovascular condition.
* Ability to provide informed consent.
* Proficient in the English language.
* Access to a device capable of running mobile application.
* Used mobile technology within the past 3 months.

Exclusion Criteria:

* Any medical condition making 1-month survival unlikely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited via emergency room (ER) visits, cardiac care unit (CCU) visits, and cardiac rehabilitation visits for any cardiac health problem over the course of the study. Cardiac conditions include the following:
  1. Atrial Fibrillation (AF).
  2. Atrial Flutter.
  3. Prior Myocardial Infarction (Post MI).
  4. Prior Coronary Artery Disease (CAD).
  5. Prosthetic Heart Valve.
  6. Dilated Aorta.
  7. Carotid Artery Disease.
  8. Peripheral Artery Disease.
  9. Diabetes Mellitus (DM).
  10. Hyperlipidemia (HLP).
  11. Hypertension (HTN).
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient Application Utilization (success is treated as ≥80% on each of the sub-items). | 1-Month.
  % of patients who completed all tasks (i.e., blood pressure entry) required of their module, % of patients who completed all 3 surveys (baseline, mid-VIRTUES, post-VIRTUES), % of patients who viewed all educational material presented to them for their module, and number of interactions with VIRTUES per week across the month.
Patient Access to Care (success is treated as ≥80% on each of the sub-items). | 1-Month.
  % of patients who self-report that the program facilitated their access to care and % of patients who self-report that the program created a higher quality of care for them.
Patient Autonomy (success is treated as ≥80%). | 1-Month.
  % of patients who self-report that the program provided them with a greater sense of autonomy in their care.
Patient Recommendation Adherence (success is treated as ≥80%). | 1-Month.
  % of patients who self-report that they have reviewed all guideline-directed recommendations given to them for their module with their healthcare provider.
Patient Overall Satisfaction (success is treated as ≥80%). | 1-Month.
  % of patients who self-report that they are overall moderately to highly satisfied with the VIRTUES program.
Qualitative Outcomes from Focus Groups. | 1-Month.
  Emerging themes on VIRTUES features to improve and modify.

SECONDARY OUTCOMES:
Physician Adherence to Guideline-Directed Recommendations (success is treated as ≥80%). | 1-Month.
  % of physicians who adhere to the recommendations.
Patient Self-Reported Improvements in Parameters Specific to Each Module's Condition (success is treated as ≥80%). | 1-Month.
  % of patients who self-report an improvement in the condition specific to their module.

OTHER OUTCOMES:
VIRTUES Application Reliability (for all reliability outcomes, success is treated as ≤20% disruptions or technical support requests). | 1-Month
  % of system disruptions over the 1-month trial use period and % of technical support requests over the 1-month trial use period.
Number of Adverse Events | 1-Month.
  % of patients who experience an adverse event that is related to their participation.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Tang, MD FRCPC, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada